CLINICAL TRIAL: NCT04353362
Title: Comparison of Ofloxacin and Metronidazole/Amoxicillin on the Treatment of Periodontitis.
Brief Title: Alternative Antibiotic Regimen in Periodontitis Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Begum Alkan, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Istanbul Medipol
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Amoxicillin; Metronidazole; Ofloxacin; Periodontitis; Root Planing
MeSH Terms: conditions — Periodontitis | interventions — Ofloxacin; Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ofloxacin group (Experimental)
  Interventions: Drug: Ofloxacin
- Amoxicillin plus Metronidazole group (Active Comparator)
  Interventions: Drug: Amoxicillin; Drug: Metronidazole

INTERVENTIONS:
Drug: Ofloxacin — 400 mg, 1 time per day for 5 days
  Arms: Ofloxacin group
Drug: Amoxicillin — 500 mg, 3 times per day for 7 days
  Arms: Amoxicillin plus Metronidazole group
Drug: Metronidazole — 500 mg, 3 times per day, for 7 days
  Arms: Amoxicillin plus Metronidazole group

SUMMARY:
Context and Aims: Several studies have demonstrated an association between obesity, periodontitis, and exercise. This study aimed to investigate the effects of regular exercise on obese women with periodontal disease, using serum, saliva, and gingival crevicular fluid (GCF) samples.

Settings and Design: A before-after study design was adopted to evaluate the effects of 12 weeks of regular exercise on obese women grouped according to periodontal status, without a control group (no exercise).

Methods and Material: The study sample comprised fifteen patients without periodontitis (NP group) and 10 patients with chronic periodontitis (CP group), from whom periodontal parameters were measured and serum, saliva, and GCF samples were collected. Body mass index (BMI), anthropometric measurements, somatotype-motoric tests, and maximal oxygen consumption (VO2max) were recorded at baseline and after exercise.

Statistical analysis used: MedCalc was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* The periodontal diagnosis of participants with generalized periodontitis stage III-IV/grade C. Systemically healthy participants with generalized periodontitis were enrolled if they were between 18 and 40 years of age, and had no allergies to penicillin, metronidazole or quinolones, a history of antibiotic therapy or periodontal therapy within the preceding six months

Exclusion Criteria:

* Subjects were excluded if they had any known systemic diseases or conditions that can/could influence the periodontal status, allergies to quinolones, penicillin or metronidazole, a history of antibiotic therapy, or periodontal treatment within the preceding six months

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Probing depth | 6-months
  Probing depth was recorded at the baseline, first, third, and sixth month. The changes were evaluated among and between groups.

SECONDARY OUTCOMES:
Clinical attachment loss | 6-months
  Clinical attachment loss was recorded at the baseline, first, third, and sixth month. The changes were evaluated among and between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Begum Alkan, Istanbul, Turkey (Türkiye)